CLINICAL TRIAL: NCT00583934
Title: Is Screening for Esophageal Pathology in Asymptomatic Patients Post-Treatment for Head and Neck Cancer Beneficial?
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Gregory Farwell, MD, University of California, Davis
Other Study IDs: 200513668-3; 00004557
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-07

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer, head and neck cancer, dysplasia
MeSH Terms: conditions — Esophageal Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Those six months post treatment for head and neck cancer.

SUMMARY:
The purpose of this study is to evaluate the prevalence of esophageal pathology in asymptomatic patients with a history of head and neck cancer.

DETAILED DESCRIPTION:
There are certain factors (i.e. alcohol, tobacco, decreased saliva production from radiation) that predispose patients with a history of head and neck cancer to have esophageal disease. Often, in the initial stages of the disease, patients do not have symptoms. However, the early detection of precancerous lesions or small cancers improves patients' chances of being cured. There is no direct data supporting the practice of screening patients with a history of head and neck cancer after treatment for esophageal disease if they are not experiencing symptoms. However, many argue that screening endoscopy is justified in high risk patients to detect early esophageal cancer or dysplasia at a curable state. We are, therefore, performing this study to determine the value of endoscopic screening of the esophagus after treatment for head and neck cancer in patients without symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer patients that are six months post treatment and asymptomatic for esophageal disease.

Exclusion Criteria:

* None if meets the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject population will be recruited from the clinical practice of the investigators.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2007-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Early detection of esophageal cancer or dysplasia in patients without symptoms, after treating their primary cancer, may improve their chances of being cured of a secondary disease.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Farwell, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States